CLINICAL TRIAL: NCT03322800
Title: A Randomised, Double-blind, Placebo-controlled, Phase I Study of Orally Administered AK0529 in Chinese Healthy Adult Volunteers
Brief Title: A Study of AK0529 to Evaluate Pharmacokinetics and Safety in Chinese Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Ark Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AK0529-2001
Record Dates: First submitted 2017-10-19; First posted 2017-10-26 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Healthy
MeSH Terms: interventions — ziresovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- AK0529 100 mg, Pilot (Experimental): This is an open pilot arm and male subjects enrolled into this arm will be only administered with an oral single dose of 100 mg AK0529. The dose group begins treatment on Day 1.
  Interventions: Drug: AK0529
- AK0529 100 mg (Experimental): Subjects will be administered with an oral single dose of 100 mg AK0529 or placebo. The dose group begins treatment on Day 1.
  Interventions: Drug: AK0529; Other: Placebo
- AK0529 300 mg, food effect (Experimental): A 3x3 cross-over study is designed in this group to evaluate the food effect following a standard Chinese meal or a high fat meal in the same subjects, comparing with the PK profile of AK0529 under fasted condition. Subjects will be administered with an oral dose of 300 mg AK0529 or placebo on Day 1 of each cycle.
  Interventions: Drug: AK0529; Other: Placebo
- AK0529 600 mg (Experimental): Subjects will be administered with an oral single dose of 600 mg AK0529 or placebo. The dose group begins treatment on Day 1.
  Interventions: Drug: AK0529; Other: Placebo
- AK0529 300 mg, MAD (Experimental): Subjects will be administered with the multiple doses of 300 mg AK0529 or placebo on Day 1-7.
  Interventions: Drug: AK0529; Other: Placebo
- Placebo (Other): For assessment of the Adverse Event (AE) profile, there are placebo controls in each dose group (except the pilot group). The placebo is administered at the same time (and of the same dosage) as the AK0529 subjects.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: AK0529 — Active Substance: AK0529, Pharmaceutical Form: Capsule, Route of Administration: Oral
  Arms: AK0529 100 mg; AK0529 100 mg, Pilot; AK0529 300 mg, MAD; AK0529 300 mg, food effect; AK0529 600 mg
Other: Placebo — Active Substance: Placebo, Pharmaceutical Form: Capsule, Route of Administration: Oral
  Arms: AK0529 100 mg; AK0529 300 mg, MAD; AK0529 300 mg, food effect; AK0529 600 mg; Placebo

SUMMARY:
This study will characterize the pharmacokinetics (PK) of AK0529, the effect of food and evaluate the safety of AK0529 in healthy Chinese adult subjects. 50 subjects will be randomized to receive a dose level of AK0529 or placebo in five groups. The total study duration will be approximately 18-27 days for each subject.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, single-center, Phase I study in healthy Chinese subjects. The objectives of the study are to evaluate the safety of AK0529, characterize the PK of AK0529 and to evaluate the effect of food in healthy Chinese subjects. 50 healthy Chinese subjects will be randomized to orally receive one of four dose levels of AK0529 (single dose:100 mg and 300 mg, Multiple dose: 600 mg, Cross-over Food Effect: 300 mg) or placebo. The total duration of the study will be approximately 18 to 27 days for each subject.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants between 18 and 45 years of age, inclusive.
* Have a body weight ≥45 kg (Female) or ≥50 kg (Male), and a body mass index (BMI) between 19 and 26 kg/m^2, inclusive.
* Participants are in good health without any significant clinical abnormalities as determined by the investigator on the basis of medical history, physical examination (including vital signs) and baseline test results (hematology, blood chemistry, blood coagulation, urinalysis and 12-lead electrocardiogram (ECG)).
* Participants and the spouses who are willing to use a medically accepted method of contraception (e.g. placement of an intrauterine device or intrauterine system, contraceptive drugs, using condom) during the study period and for one month thereafter.
* Participants who are willing to sign and date the approved informed consent form (ICF).

Exclusion Criteria:

* Female subjects of childbearing potential have positive serum pregnancy test results or are lactating at screening.
* Subjects who have their daily cigarette smoking to five or more for 3 months prior to screening.
* History of severe or multiple drug allergies.
* History of alcohol abuse in the past 3 months prior to screening (Alcohol consumption >14 units per week: 1 unit = 10 mL alcohol, 250mL of 4 degrees beer, 25 mL of 40 degrees spirit or 75 mL of 13 degrees wine).
* History of any drug abuse, or have a positive urine drug screen result at screening, or history of any psychotropic medication abuse within 5 years prior to screening.
* Previous exposure to any other Investigational Medicinal Product (IMP) or participation in any clinical trial within 3 months prior to screening.
* Donation or loss of blood over 450 mL within 3 months prior to screening.
* Use of any prescription, over-the-counter, herbs, or medications which can change the pH values of gastrointestinal tracts (e.g. antacids, H2 receptor inhibitors and/or proton-pump inhibitors) within 28 days prior to screening.
* Receiving caffeine-containing food or drinks, or alcohol-containing products within 24 hours prior to study drug administration.
* Smoking and use of any nicotine-containing products within 24 hours prior to study drug administration.
* Have swallowing problems, or any gastrointestinal diseases or history of surgery (e.g. subtotal gastrectomy) that could possibly affect drug absorption.
* Clinically relevant abnormalities in the ECG results.
* Clinically significant abnormalities in the lab test results of biochemistry, hematology, blood coagulation or urinalysis above the upper limit of normal (ULN) ranges as judged by the investigator.
* Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab), human immunodeficiency virus (HIV-1 or HIV-2 antibody) or syphilis results.
* Evidence of clinical significant digestive, urological, neurological,hematological, endocrine, oncological, pulmonary, immunological, cardiovascular, or psychiatric disease at screening.
* ECG results with the QT interval, corrected for heart rate by Bazett's formula (QTcB) of > 450 msec in the supine position at screening.
* Systolic blood pressure (SBP) > 140 mmHg or < 90 mmHg, and/or diastolic blood pressure (DBP) > 90 mmHg or < 60 mmHg in the seated position at screening.
* Subjects are lactose intolerant.
* Inability to meet the study requirements in the opinion of the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2018-04-06 (Actual); Study Completion 2018-05-24 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Day1 (pre-dose and 0.5,1,1.5,2,3,4,5,6,8,10,12 hrs post-dose), Day2 (24 hrs post-dose), Day3 (48 hrs post-dose), Day4 (72 hrs post-dose), Day5, Day6, Day7, Day8, Day9 and Day10
  The maximum observed plasma concentration of AK0529.
Time to Maximum Plasma Concentration (Tmax) | Day1 (pre-dose and 0.5,1,1.5,2,3,4,5,6,8,10,12 hrs post-dose), Day2 (24 hrs post-dose), Day3 (48 hrs post-dose), Day4 (72 hrs post-dose), Day5, Day6, Day7, Day8, Day9 and Day10
  The time of occurrence of Cmax.
Area under the plasma concentration-time curve from time zero up to time (AUC 0-t) | Day1 (pre-dose and 0.5,1,1.5,2,3,4,5,6,8,10,12 hrs post-dose), Day2 (24 hrs post-dose), Day3 (48 hrs post-dose), Day4 (72 hrs post-dose), Day5, Day6, Day7, Day8, Day9 and Day10
  The area under the plasma concentration-time curve from time zero up to the last analytically quantifiable concentration of AK0529.
Terminal Half-Life (t1/2) | Day1 (pre-dose and 0.5,1,1.5,2,3,4,5,6,8,10,12 hrs post-dose), Day2 (24 hrs post-dose), Day3 (48 hrs post-dose), Day4 (72 hrs post-dose), Day5, Day6, Day7, Day8, Day9 and Day10
  The apparent elimination half-life of AK0529.
Area Under the Plasma Concentration-Time Curve Extrapolated to Infinity (AUC0-inf) | Day1 (pre-dose and 0.5,1,1.5,2,3,4,5,6,8,10,12 hrs post-dose), Day2 (24 hrs post-dose), Day3 (48 hrs post-dose), Day4 (72 hrs post-dose), Day5, Day6, Day7, Day8, Day9 and Day10
  The area under the plasma concentration-time curve from time zero up extrapolated to infinity of AK0529.
Apparent Oral Clearance (CL/F) | Day1 (pre-dose and 0.5,1,1.5,2,3,4,5,6,8,10,12 hrs post-dose), Day2 (24 hrs post-dose), Day3 (48 hrs post-dose), Day4 (72 hrs post-dose), Day5, Day6, Day7, Day8, Day9 and Day10
  The oral clearance of AK0529
Percentage of Subjects with Adverse Events (AEs) | From baseline up to approximately 6 weeks
  An adverse event can be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product.

CONTACTS AND LOCATIONS:
Overall Officials: Jimmy Gu, Study Director — info@arkbiosciences.com
Locations (1):
- Shanghai Xuhui Central Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No